CLINICAL TRIAL: NCT06746389
Title: Effects of Vitamin D Supplementation on Myofibrillar Protein Synthesis Rates in Rested and Exercised Muscle in Young Adults: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Effects of Vitamin D Supplementation on Muscle Protein Synthesis
Acronym: VIPER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other); Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201021/B/03
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Vitamin D Effects on MPS; Placebo Effects on MPS
Keywords: Muscle Protein Synthesis, Vitamin D, adults, healthy

STUDY DESIGN:
Intervention Model Description: Double Blind RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Experimental): 3000 IU/Day 12 weeks
  Interventions: Dietary Supplement: 3000 IU per Day Spray
- Placebo (Placebo Comparator): Placebo one/day 12 weeks
  Interventions: Dietary Supplement: 3000 IU per Day Spray

INTERVENTIONS:
Dietary Supplement: 3000 IU per Day Spray — Effects of vitamin D supplementation vs placebo on MPS in response to exercise and feeding

SUMMARY:
Background: Healthy adults maintain muscle tissue by continuously building up and breaking down muscle proteins throughout the day. Studies have shown that vitamin D (VitD) is essential for maintaining muscle mass by activating cellular pathways involved in building muscle via muscle protein synthesis (MPS). Although, various candidate molecules have been identified in animal models, it is not known whether these pathways are activated in humans. Interestingly, animal studies indicate that 20% of VitD is stored in human muscle cells, which may help maintain VitD sufficiency during winter in Northern latitudes when there is not much sunlight Objectives: We will investigate whether VitD supplementation increases the MPS response to feeding and exercise, VitD storage in muscle cells, and cellular pathways that are involved in healthy sedentary or moderately active adults.

Methods: Participants will consume either a placebo (sucrose) or the intervention (vitamin D3, 3000IU/day) for 12 weeks in a double-blinded randomised study. Before and after the intervention participants will have body composition measured. Blood and muscle samples will be taken before and after a bout of exercise and ingestion of 20 g protein in order to measure MPS.

DETAILED DESCRIPTION:
Recent in vitro studies have demonstrated an anabolic role of vitamin D directly targeting skeletal muscle via vitamin D receptors (VDR) present in myotubes [1,2,3]. However, this has yet to be translated to in vivo human models.

25-hydroxyvitamin-D (25OHD) is the primary circulating metabolite and reference measurement for vitamin D status. This may then either be converted to 24,25-dihydroxyvitamin D3 (24,25OHD) to prevent intoxication [4] or be activated in the kidneys to 1,25-dihydroxyvitamin D (1,25OHD)[5].

Evidence support a biological role for 1,25OHD in skeletal muscle[1-4,7]. With focus on muscle hypertrophy, a study demonstrated that 25OHD can also be activated to 1,25OHD in myotubes[8] and promote cell proliferation, growth and differentiation of myocytes in in vitro skeletal muscle cells[7,9-13]. The mechanisms proposed include (i) gene expression of endocytic receptors for vitamin D binding protein (VDP) (megalin/cubulin) on the muscle cell surface membrane and (ii) high affinity for VDP to bind to actin inside the muscle cell. Furthermore, epidemiological studies support a positive role for vitamin D in human muscle function[14-21] and mechanistic studies implicate intracellular 25OHD in the regulation of protein metabolism. Cell culture and in vivo animal models demonstrate that 25OHD activates anabolic cell signalling proteins of the mTORC1 pathway in response to anabolic stimuli[21,22], which translates into an increased stimulation of muscle protein synthesis[17]. Despite these exciting results from cell culture and in vivo animal studies, no study has replicated these findings in in vivo human models.

The length of the intervention in studies investigating the effects of vitamin D supplementation on muscle health outcomes and MPS varies between studies; however, evidence supports improvements in fast-twitch muscle fibres in elderly women[18], muscle strength in humans and animals and an increased in MPS in rats and mice following a minimum of 12 weeks intervention [22]. Thus, this study plans to have 12 weeks of intervention to ensure there is sufficient time for a physiologically effect to take place. Seasonal variations in blood 25OHD concentrations have been evaluated in Caucasians residing in Northern Ireland[4]. Thirty-four percent were deficient (<25nmol/L) in winter months[4]; however, despite insufficient sunlight in winter to synthesise vitamin D in skin, a significant proportion of a population resident in the same latitude, in Scotland, maintained blood 25OHD concentrations >50nmol/L[6]. These data and a recent review[8] suggest that humans have evolved a storage mechanism, which allows 25OHD, produced in the summer, to be conserved and used more efficiently in winter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 - 45
* Sedentary and moderately active (NDNS)

Exclusion Criteria:

* Any diagnosed acute or chronic condition
* Very active (NDNS)
* On medication apart from contraceptive pill
* Not taking vitamin supplementation for 30 days before enrolling
* Not having been exposed to the sun (synthesising months - any country) in the previous 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Any
Enrollment: 18 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate of amino acid incorporation into myofibrillar protein | 12 weeks x 4 time points
  Fractional synthetic rate of amino acid incorporation into myofibrillar protein

SECONDARY OUTCOMES:
Phosphorylated mTOR | 12 weeks x 4 time points
  Phosphorylated mTOR response following 12 weeks intervention vs placebo
Total mTOR | 12 weeks x 2 time points
  Total mTOR following 12 weeks intervention
Plasma amino acid kinetics | 12 weeks x 16 time points
  Plasma amino acid kinetics in response to intervention vs. placebo
Glucose | 12 weeks x 16 time points
  Glucose response to intervention vs. placebo
Insulin | 12 weeks x 14 time points
  Insulin response to intervention vs. placebo
Leg press | 12 weeks x 1 x1
  Leg press - strength
Leg extension | 12 weeks 1 x 1
  Leg extension - Strength

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Revuelta Iniesta, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to data protection - participants did not agree to IPD

REFERENCES:
- [Background] Tieland M, Brouwer-Brolsma EM, Nienaber-Rousseau C, van Loon LJ, De Groot LC. Low vitamin D status is associated with reduced muscle mass and impaired physical performance in frail elderly people. Eur J Clin Nutr. 2013 Oct;67(10):1050-5. doi: 10.1038/ejcn.2013.144. Epub 2013 Aug 14. PMID 23942175
- [Background] Vignale K, Greene ES, Caldas JV, England JA, Boonsinchai N, Sodsee P, Pollock ED, Dridi S, Coon CN. 25-Hydroxycholecalciferol Enhances Male Broiler Breast Meat Yield through the mTOR Pathway. J Nutr. 2015 May;145(5):855-63. doi: 10.3945/jn.114.207936. Epub 2015 Mar 18. PMID 25788584
- [Background] Salles J, Chanet A, Giraudet C, Patrac V, Pierre P, Jourdan M, Luiking YC, Verlaan S, Migne C, Boirie Y, Walrand S. 1,25(OH)2-vitamin D3 enhances the stimulating effect of leucine and insulin on protein synthesis rate through Akt/PKB and mTOR mediated pathways in murine C2C12 skeletal myotubes. Mol Nutr Food Res. 2013 Dec;57(12):2137-46. doi: 10.1002/mnfr.201300074. Epub 2013 Aug 9. PMID 23929734
- [Background] Chiang CM, Ismaeel A, Griffis RB, Weems S. Effects of Vitamin D Supplementation on Muscle Strength in Athletes: A Systematic Review. J Strength Cond Res. 2017 Feb;31(2):566-574. doi: 10.1519/JSC.0000000000001518. PMID 27379960
- [Background] Beals JW, Sukiennik RA, Nallabelli J, Emmons RS, van Vliet S, Young JR, Ulanov AV, Li Z, Paluska SA, De Lisio M, Burd NA. Anabolic sensitivity of postprandial muscle protein synthesis to the ingestion of a protein-dense food is reduced in overweight and obese young adults. Am J Clin Nutr. 2016 Oct;104(4):1014-1022. doi: 10.3945/ajcn.116.130385. Epub 2016 Sep 7. PMID 27604771
- [Background] Montenegro KR, Cruzat V, Carlessi R, Newsholme P. Mechanisms of vitamin D action in skeletal muscle. Nutr Res Rev. 2019 Dec;32(2):192-204. doi: 10.1017/S0954422419000064. Epub 2019 Jun 17. PMID 31203824
- [Background] van Vliet S, Fappi A, Reeds DN, Mittendorfer B. No independent or combined effects of vitamin D and conjugated linoleic acids on muscle protein synthesis in older adults: a randomized, double-blind, placebo-controlled clinical trial. Am J Clin Nutr. 2020 Nov 11;112(5):1382-1389. doi: 10.1093/ajcn/nqaa240. PMID 32860399
- [Background] Holick MF. High prevalence of vitamin D inadequacy and implications for health. Mayo Clin Proc. 2006 Mar;81(3):353-73. doi: 10.4065/81.3.353. PMID 16529140
- [Background] SANC. (2007) Update on Vitamin D: Position Statement by the Scientific Advisory Committee on Nutrition. London: TSO
- [Background] Mann CJ, Perdiguero E, Kharraz Y, Aguilar S, Pessina P, Serrano AL, Munoz-Canoves P. Aberrant repair and fibrosis development in skeletal muscle. Skelet Muscle. 2011 May 4;1(1):21. doi: 10.1186/2044-5040-1-21. PMID 21798099
- [Background] Relaix F, Zammit PS. Satellite cells are essential for skeletal muscle regeneration: the cell on the edge returns centre stage. Development. 2012 Aug;139(16):2845-56. doi: 10.1242/dev.069088. PMID 22833472
- [Background] Owens DJ, Sharples AP, Polydorou I, Alwan N, Donovan T, Tang J, Fraser WD, Cooper RG, Morton JP, Stewart C, Close GL. A systems-based investigation into vitamin D and skeletal muscle repair, regeneration, and hypertrophy. Am J Physiol Endocrinol Metab. 2015 Dec 15;309(12):E1019-31. doi: 10.1152/ajpendo.00375.2015. Epub 2015 Oct 27. PMID 26506852
- See also: The overarching aim of this project is to investigate if vitamin D supplementation can increase muscle mass and strength and to explore if the cellular pathways identified in healthy individuals — https://medicine.exeter.ac.uk/phss/research/foodnutrition/clinical/
- Available data/document: Protocol and ethics can be shared on request: 201021/B/03 — https://www.exeter.ac.uk/departments/cgr/researchethics/ — Ethics documents and study protocol can be shared on request. Please contact PI Dr Raquel Revuelta Iniesta at r.revuelta-iniesta@exeter.ac.uk or the PHSS Ethics Committee at a.guy@exeter.ac.uk